CLINICAL TRIAL: NCT01833026
Title: Comparative Effectiveness of COPD Assessment and Management Bundle Versus Usual Care in Patients Suspected of Having COPD
Brief Title: COPD Assessment and Management Bundle Versus Usual Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Min Joo, MD MPH, Assistant Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012-0997; K23HL094461 (NIH)
Record Dates: First submitted 2013-04-11; First posted 2013-04-16 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: pulmonary disease; chronic obstructive airflow; spirometry; primary healthcare; guideline-based therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — Spirometry; Levalbuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COPD assessment and management recommendations (Experimental): Patients with a physician-diagnosed COPD or asthma suspicious for COPD being managed by the physician randomized to the intervention group will perform a spirometry test and provide information regarding their medical history on their initial visit, which is 90 minutes before their doctor's appointment. A letter containing the interpretation of spirometry test results, and recommendations for guideline based therapy based on GOLD guidelines will be available to the primary care doctor at the time of the patient's clinic visit. The doctor may review the results and use his or her own judgment in moving forward with the subject's diagnosis and management. A copy of the spirometry results and assessment based on the GOLD criteria at the time of the test of your subject will be uploaded to his or her electronic health record for future reference.
  Outcomes will be assessed every 3 months for up to one year through patient telephone calls and medical chart reviews.
  Interventions: Device: Spirometry test; Drug: Levalbuterol
- Usual Care (Placebo Comparator): Patients with a physician-diagnosed COPD or physician-diagnosed asthma suspicious for COPD being managed by the physician randomized to the usual care group will provide medical history, not initially have a spirometry, and will be observed as usual care.
  Outcomes will be assessed every 3 months for up to one year through patient telephone calls and medical chart reviews. At the conclusion of the research study which will be 12 months from the patients' initial visit, patients being managed by the physician randomized to the usual care group will have a spirometry test and these results will not be shared with the doctor or the patients during the study but will be uploaded to the electronic health record after the end of the study for future reference.
  Interventions: Device: Spirometry test; Drug: Levalbuterol

INTERVENTIONS:
Device: Spirometry test — For the initial visit for the intervention group, an initial demographics form and a health questionnaire will given to the subject to complete. To evaluate the breathing and quality of living, a spirometry test will be performed that will evaluate how well and how fast the subject can breath and blow out air.
  Other Names: KoKo Spirometer (Model 313105); 3 Liter Calibration Syringe
Drug: Levalbuterol — The spirometry test will be performed with a breathing medication called Levalbuterol (Xopenex®). Levalbuterol is used in standard practice for COPD and is commonly used during spirometry.
  Other Names: Xopenex®: 4 puffs administered 30 seconds apart

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a progressive respiratory (lung) disease that makes it harder to breathe over time. To date, there is no cure for COPD, but it can be managed when diagnosed and proper medical care is provided.

The purpose of this study is to determine if diagnosis and guided therapy with the use of spirometry is related to better patient outcomes (the condition of a patient's health) compared to usual care which may or may not include the use of spirometry. Spirometry is a standardized test used in medical practice that measures how much air your lungs can hold and how forcefully you can breathe out.

For this study, the investigators will compare two groups: 1) intervention (treatment) group and 2) usual care group (control). The intervention group will have a spirometry test and the results will be provided to the primary care physician. The usual care group will not initially have a spirometry test. Both groups will be followed for outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to determine if diagnosis and guided therapy with the use of spirometry is related to better patient associated outcomes compared to usual care which may or may not include the use of spirometry. To do this, we propose a comparative effectiveness trial of introducing a COPD assessment and management bundle targeted to primary care providers for patients suspected of having COPD versus usual care.

ELIGIBILITY:
Inclusion Criteria:

Patients, male and female, who are at least 40 years of age, receive primary treatment at the University of Illinois , and with any one of the following:

New Diagnosis

Inpatient or emergency department setting

1. New physician-diagnosis of COPD and/or new physician-diagnosis of asthma with a ≥10 pack year smoking without a spirometry 4 weeks or more after discharge from diagnosis setting.

   Outpatient setting
2. A new physician diagnosis of COPD within the past 6 months prior to their visit, without a spirometry or with a normal spirometry within the past 5 years prior to the diagnosis to the time of their visit.
3. A new physician diagnosis of asthma within past 6 months and a ≥10 pack year smoking history prior to their visit, without a diagnosis of COPD, without a spirometry or with a pre-bronchodilator spirometry with evidence of obstruction within the past 5 years prior to the diagnosis to the time of their visit.
4. Any patient with an existing physician-diagnosis of asthma within the past 2 years but > 6 months prior to the time of their visit and a ≥10 pack year smoking history, without a diagnosis of COPD, using a respiratory medication in the past year, and no spirometry on record or had a pre-bronchodilator spirometry with evidence of obstruction on record for at least the past 5 years.

   Existing Diagnosis
5. Any patient with an existing physician-diagnosis of COPD within the past 2 years but > 6 months prior to the time of their visit, and using a respiratory medication in the past year but no spirometry on record or had a spirometry without evidence of chronic obstruction in the past 5 years.

Exclusion Criteria:

1. Unable to perform adequate spirometry (e.g. muscle weakness, tracheostomy, cognitive dysfunction, mental retardation or other psychiatric disorders)
2. Non-English speaking
3. Pregnancy
4. Any patient planning to move away from the city within the next year.
5. Seen by a pulmonary specialist in the past 3 years.
6. Any terminal illness with a life expectancy of <6 months (e.g. hospice care, malignancies)
7. Any patient with a physician diagnosis of COPD and had a pre or post-bronchodilator spirometry with evidence of chronic obstruction on record.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Joo, MD, MPH, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois, Chicago, Illinois, United States

REFERENCES:
- [Background] Global Initiative for Chronic Obstructive Lung Disease. Global strategy for the diagnosis, management and prevention of chronic obstructive pulmonary disease: World Health Organization and National Heart, Lung, and Blood Institute, 2011
- [Background] Akinbami LJ, Liu X. Chronic obstructive pulmonary disease among adults aged 18 and over in the United States, 1998-2009. NCHS Data Brief. 2011 Jun;(63):1-8. PMID 22142836
- [Background] Sullivan SD, Ramsey SD, Lee TA. The economic burden of COPD. Chest. 2000 Feb;117(2 Suppl):5S-9S. doi: 10.1378/chest.117.2_suppl.5s. PMID 10673466
- [Background] Mapel DW, Hurley JS, Frost FJ, Petersen HV, Picchi MA, Coultas DB. Health care utilization in chronic obstructive pulmonary disease. A case-control study in a health maintenance organization. Arch Intern Med. 2000 Sep 25;160(17):2653-8. doi: 10.1001/archinte.160.17.2653. PMID 10999980
- [Background] Chronic obstructive pulmonary disease data fact sheet: U.S. Department of Health and Human Services, National Institutes of Health, National Heart, Lung and Blood Institute, 2003
- [Background] Morbidity and mortality: 2009 chartbook on cardiovascular, lung and blood diseases: National Heart Lung and Blood Institute, 2009
- [Background] Han MK, Kim MG, Mardon R, Renner P, Sullivan S, Diette GB, Martinez FJ. Spirometry utilization for COPD: how do we measure up? Chest. 2007 Aug;132(2):403-9. doi: 10.1378/chest.06-2846. Epub 2007 Jun 5. PMID 17550936
- [Background] Joo MJ, Lee TA, Weiss KB. Geographic variation of spirometry use in newly diagnosed COPD. Chest. 2008 Jul;134(1):38-45. doi: 10.1378/chest.08-0013. Epub 2008 Mar 17. PMID 18347201
- [Background] Lee TA, Bartle B, Weiss KB. Spirometry use in clinical practice following diagnosis of COPD. Chest. 2006 Jun;129(6):1509-15. doi: 10.1378/chest.129.6.1509. PMID 16778268
- [Background] Damarla M, Celli BR, Mullerova HX, Pinto-Plata VM. Discrepancy in the use of confirmatory tests in patients hospitalized with the diagnosis of chronic obstructive pulmonary disease or congestive heart failure. Respir Care. 2006 Oct;51(10):1120-4. PMID 17005056
- [Background] Joo MJ, Au DH, Fitzgibbon ML, McKell J, Lee TA. Determinants of spirometry use and accuracy of COPD diagnosis in primary care. J Gen Intern Med. 2011 Nov;26(11):1272-7. doi: 10.1007/s11606-011-1770-1. Epub 2011 Jun 29. PMID 21713542
- [Background] Badgett RG, Tanaka DJ, Hunt DK, Jelley MJ, Feinberg LE, Steiner JF, Petty TL. The clinical evaluation for diagnosing obstructive airways disease in high-risk patients. Chest. 1994 Nov;106(5):1427-31. doi: 10.1378/chest.106.5.1427. PMID 7956395
- [Background] Buffels J, Degryse J, Heyrman J, Decramer M; DIDASCO Study. Office spirometry significantly improves early detection of COPD in general practice: the DIDASCO Study. Chest. 2004 Apr;125(4):1394-9. doi: 10.1378/chest.125.4.1394. PMID 15078751
- [Background] Straus SE, McAlister FA, Sackett DL, Deeks JJ; CARE-COAD2 Group. Clinical Assessment of the Reliability of the Examination-Chronic Obstructive Airways Disease. Accuracy of history, wheezing, and forced expiratory time in the diagnosis of chronic obstructive pulmonary disease. J Gen Intern Med. 2002 Sep;17(9):684-8. doi: 10.1046/j.1525-1497.2002.20102.x. PMID 12220364
- [Background] van Schayck CP, van Weel C, Harbers HJ, van Herwaarden CL. Do physical signs reflect the degree of airflow obstruction in patients with asthma or chronic obstructive pulmonary disease? Scand J Prim Health Care. 1991 Dec;9(4):232-8. doi: 10.3109/02813439109018525. PMID 1792447
- [Background] Straus SE, McAlister FA, Sackett DL, Deeks JJ. The accuracy of patient history, wheezing, and laryngeal measurements in diagnosing obstructive airway disease. CARE-COAD1 Group. Clinical Assessment of the Reliability of the Examination-Chronic Obstructive Airways Disease. JAMA. 2000 Apr 12;283(14):1853-7. doi: 10.1001/jama.283.14.1853. PMID 10770147
- [Background] Holleman DR Jr, Simel DL. Does the clinical examination predict airflow limitation? JAMA. 1995 Jan 25;273(4):313-9. No abstract available. PMID 7815660
- [Background] Bolton CE, Ionescu AA, Edwards PH, Faulkner TA, Edwards SM, Shale DJ. Attaining a correct diagnosis of COPD in general practice. Respir Med. 2005 Apr;99(4):493-500. doi: 10.1016/j.rmed.2004.09.015. Epub 2004 Nov 11. PMID 15763457
- [Background] Mannino DM, Homa DM, Akinbami LJ, Ford ES, Redd SC. Chronic obstructive pulmonary disease surveillance--United States, 1971-2000. MMWR Surveill Summ. 2002 Aug 2;51(6):1-16. PMID 12198919
- [Background] Mannino DM, Gagnon RC, Petty TL, Lydick E. Obstructive lung disease and low lung function in adults in the United States: data from the National Health and Nutrition Examination Survey, 1988-1994. Arch Intern Med. 2000 Jun 12;160(11):1683-9. doi: 10.1001/archinte.160.11.1683. PMID 10847262
- [Background] Tinkelman DG, Price DB, Nordyke RJ, Halbert RJ. Misdiagnosis of COPD and asthma in primary care patients 40 years of age and over. J Asthma. 2006 Jan-Feb;43(1):75-80. doi: 10.1080/02770900500448738. PMID 16448970
- [Background] Walker PP, Mitchell P, Diamantea F, Warburton CJ, Davies L. Effect of primary-care spirometry on the diagnosis and management of COPD. Eur Respir J. 2006 Nov;28(5):945-52. doi: 10.1183/09031936.06.00019306. Epub 2006 Jul 26. PMID 16870668
- [Background] Mapel DW, Dutro MP, Marton JP, Woodruff K, Make B. Identifying and characterizing COPD patients in US managed care. A retrospective, cross-sectional analysis of administrative claims data. BMC Health Serv Res. 2011 Feb 23;11:43. doi: 10.1186/1472-6963-11-43. PMID 21345188
- [Background] Schnell K, Weiss CO, Lee T, Krishnan JA, Leff B, Wolff JL, Boyd C. The prevalence of clinically-relevant comorbid conditions in patients with physician-diagnosed COPD: a cross-sectional study using data from NHANES 1999-2008. BMC Pulm Med. 2012 Jul 9;12:26. doi: 10.1186/1471-2466-12-26. PMID 22695054
- [Background] Calverley PM, Anderson JA, Celli B, Ferguson GT, Jenkins C, Jones PW, Yates JC, Vestbo J; TORCH investigators. Salmeterol and fluticasone propionate and survival in chronic obstructive pulmonary disease. N Engl J Med. 2007 Feb 22;356(8):775-89. doi: 10.1056/NEJMoa063070. PMID 17314337
- [Background] Ernst P, Gonzalez AV, Brassard P, Suissa S. Inhaled corticosteroid use in chronic obstructive pulmonary disease and the risk of hospitalization for pneumonia. Am J Respir Crit Care Med. 2007 Jul 15;176(2):162-6. doi: 10.1164/rccm.200611-1630OC. Epub 2007 Mar 30. PMID 17400730
- [Background] Kardos P, Wencker M, Glaab T, Vogelmeier C. Impact of salmeterol/fluticasone propionate versus salmeterol on exacerbations in severe chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2007 Jan 15;175(2):144-9. doi: 10.1164/rccm.200602-244OC. Epub 2006 Oct 19. PMID 17053207
- [Background] Lee TA, Pickard AS, Au DH, Bartle B, Weiss KB. Risk for death associated with medications for recently diagnosed chronic obstructive pulmonary disease. Ann Intern Med. 2008 Sep 16;149(6):380-90. doi: 10.7326/0003-4819-149-6-200809160-00004. PMID 18794557
- [Background] Singh S, Loke YK, Furberg CD. Inhaled anticholinergics and risk of major adverse cardiovascular events in patients with chronic obstructive pulmonary disease: a systematic review and meta-analysis. JAMA. 2008 Sep 24;300(12):1439-50. doi: 10.1001/jama.300.12.1439. PMID 18812535

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: None to report
Groups:
- Intervention: Patients with a physician-diagnosed COPD or physician-diagnosed asthma suspicious for COPD being managed by the physician randomized to the usual care group will provide medical history, not initially have a spirometry, and will be observed as usual care.
  Outcomes will be assessed every 3 months for up to one year through patient telephone calls and medical chart reviews. At the conclusion of the research study which will be 12 months from the patients' initial visit, patients being managed by the physician randomized to the usual care group will have a spirometry test and these results will not be shared with the doctor or the patients during the study but will be uploaded to the electronic health record after the end of the study for future reference.
  Spirometry test: For the initial visit for the intervention group, an initial demographics form and a health questionnaire will given to the subject to complete. To evaluate the breathing and quality of living, a spirometry test
Period: Overall Study
Arm/Group | Usual Care | Intervention
Started | 22 | 34
Completed | 22 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COPD Assessment and Management Recommendations | Usual Care | Total
Number analyzed (Participants) | 34 | 22 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 13 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.1) | 57.0 (6.9) | 58.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 39
  Male | 12 | 5 | 17
Region of Enrollment [Number; unit: participants]
  United States | 34 | 22 | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Accurate Classification of Irreversible Airflow Obstruction
Description: accuracy of diagnosis was the outcome measure. The results of the spirometry test (done in the beginning for the intervention group and ant the end of 1 year for the usual care groups) were reviewed in conjunction with the initial physician diagnosis of COPD and/or asthma to confirm whether the diagnosis was accurate, not accurate, or indeterminate. Accuracy of diagnosis of COPD was determined by spirometry results if the FEV1/FVC ratio was <0.7.
Time Frame: spirometry was performed at the first visit for intervention group and at 1 year from recruitment for the usual care group, one time assessment for both groups
Measure: Count of Participants; unit: Participants
Arm/Group | COPD Assessment and Management Recommendations | Usual Care
Number analyzed (Participants) | 34 | 22
Participants | 10 | 5

ADVERSE EVENTS:
Arm/Group | COPD Assessment and Management Recommendations | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/22
Other Adverse Events (participants affected / at risk) | 0/34 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No